CLINICAL TRIAL: NCT00266695
Title: Open-Label Treatment for Patients Completing Study B7A-MC-MBCM
Brief Title: Treatment for Completers of the Study B7A-MC-MBCM
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Chromaderm, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 10699; B7A-MC-MBDV (Other: Eli Lilly and Company)
Record Dates: First submitted 2005-12-15; First posted 2005-12-19 (Estimated); Results first posted 2016-01-28 (Estimated); Last update posted 2016-10-06 (Estimated); Status verified 2016-08

CONDITIONS: Diabetic Retinopathy
MeSH Terms: conditions — Diabetic Retinopathy | interventions — ruboxistaurin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Ruboxistaurin (Experimental)
  Interventions: Drug: Ruboxistaurin

INTERVENTIONS:
Drug: Ruboxistaurin — 32-milligram (mg) tablet, orally, once daily (QD) for up to 2 years.
  Other Names: LY 333531; Arxxant

SUMMARY:
To provide ruboxistaurin treatment to patients who completed the B7A-MC-MBCM study (NCT00604383), and who are felt by the investigator to have the potential to benefit from the ruboxistaurin treatment. Patients must be off study drug for 6 to 18 months from completion of B7A-MC-MBCM before beginning B7A-MC-MBDV. Additional data will be gathered to determine the long-term safety and effect of ruboxistaurin on vision.

ELIGIBILITY:
Inclusion Criteria:

* Patients that completed Month 36 (Visit 15) of the study B7A-MC-MBCM, and the investigator believes he/she would benefit from ruboxistaurin treatment.

Exclusion Criteria:

* Patients that discontinued from the study B7A-MC-MBCM and/or the investigator does not believe he/she would benefit from ruboxistaurin treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 203 (Actual)
Dates: Start 2006-01; Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Karl Beutner, Study Director — Chromaderm, Inc.
Locations (29):
- United States (29):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician. test, Mesa, Arizona
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician. test, Phoenix, Arizona
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician. test, Huntington Beach, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician. test, Orange, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician. test, Sacramento, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician. test, Hamden, Connecticut
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician. test, Newark, Delaware
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician. test, Tampa, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician. test, Honolulu, Hawaii
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician. test, Wheaton, Illinois
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician. test, Indianapolis, Indiana
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician. test, Shawnee Mission, Kansas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician. test, Baltimore, Maryland
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician. test, Towson, Maryland
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician. test, Boston, Massachusetts
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician. test, Grand Rapids, Michigan
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician. test, Royal Oak, Michigan
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician. test, Columbia, Missouri
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician. test, Staten Island, New York
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician. test, Charlotte, North Carolina
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician. test, Beachwood, Ohio
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician. test, Cincinnati, Ohio
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician. test, Hershey, Pennsylvania
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician. test, Pittsburgh, Pennsylvania
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician. test, Columbia, South Carolina
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician. test, Rapid City, South Dakota
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician. test, Dallas, Texas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician. test, Salt Lake City, Utah
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician. test, Madison, Wisconsin

REFERENCES:
- See also: Lilly Clinical Trial Registry — http://lillytrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study, B7A-MC-MBDV (MBDV), was an open-label extension of Study B7A-MC-MBCM (MBCM; NCT00604383), and was only open to participants who completed Study MBCM. Unless otherwise stated, the time frames refer to this study, MBDV.
Groups:
- Ruboxistaurin: 32 milligrams (mg) given once daily as an oral tablet for 2 years.
Period: Overall Study
Arm/Group | Ruboxistaurin
Started | 203
Completed | 174
Not Completed | 29
Not completed — Adverse Event | 1
Not completed — Death | 9
Not completed — Physician Decision | 1
Not completed — Lost to Follow-up | 3
Not completed — Withdrawal by Subject | 15

BASELINE CHARACTERISTICS:
Population: All enrolled participants.
Groups:
- Ruboxistaurin: 32 mg given once daily as oral tablet for 2 years.
Arm/Group | Ruboxistaurin
Number analyzed (Participants) | 203
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.50 (9.70)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 70
  Male | 133
Race/Ethnicity, Customized [Number; unit: participants]
  Caucasian | 180
  Non-Caucasian | 23
Region of Enrollment [Number; unit: participants]
  United States | 203
Diabetes Type [Number; unit: participants] — Type 1 diabetes results from autoimmune mediated destruction of the beta cells of the pancreas. Participants require insulin treatment to survive. Type 2 diabetes is characterized by resistance to the action of insulin leading to relative insulin deficiency.
  participants
    Type 1 | 24
    Type 2 | 179
Duration of Diabetes [Mean (Standard Deviation); unit: years] | 16.08 (8.40)
Body Mass Index [Mean (Standard Deviation); unit: kilograms per square meter (kg/m^2)] — Body mass index was an estimate of body fat based on body weight divided by height squared.
  kilograms per square meter (kg/m^2) | 33.47 (7.34)
Number of Diabetic Retinopathy (DR) Study Eyes Per Participant [Number; unit: participant]
  One | 72
  Two | 131
Visual Acuity (VA) Score [Mean (Standard Deviation); unit: letters read correctly] — Best-corrected Early Treatment of Diabetic Retinopathy Study (ETDRS) VA was measured at 4 meters (m) using an eye chart, 5 letters per row. Participants read chart from top down until reaching row where ≥3 letters not read correctly. If <20 letters read correctly at 4 m, chart was re-read at 1 m. Best-corrected ETDRS VA score was the total number of letters read correctly at 4 m, and if necessary, 1 m. A correction factor of 30 was added to score if total number of letters read correctly at 4 m was ≥20. VA scores ranged from 0 (no letters read correctly) to 100 (all letters read correctly).
  letters read correctly | 76.84 (13.11)
Blood Pressure [Mean (Standard Deviation); unit: millimeters of mercury (mm Hg)]
  Systolic Blood Pressure | 131.48 (17.03)
  Diastolic Blood Pressure | 73.29 (10.07)

OUTCOME MEASURES:

1. Primary Outcome: Sustained Moderate Visual Loss (SMVL)
Description: The number of participants who experienced SMVL in at least 1 diabetic retinopathy (DR) study eye. SMVL was a ≥15-letter decrease from baseline in best-corrected Early Treatment Diabetic Retinopathy Study (ETDRS) visual acuity (VA) that was sustained for the last 6 months of the study. Best-corrected ETDRS VA was measured at 4 meters (m) using an eye chart with 5 letters per row of decreasing letter size in each successive row. Participants read the chart from the top down until reaching a row where ≥3 letters in the row could not be read correctly. If <20 letters were read correctly at 4 m, the chart was re-read at 1 m. The best-corrected ETDRS VA score was the total number of letters read correctly per eye at 4 m, plus a correction factor of 30 if ≥20 letters were read correctly at 4 m, plus the total number of letters read correctly at 1 m, if assessed. Best-corrected ETDRS VA scores ranged from 0 (no letters read correctly) to 100 (all letters read correctly).
Time Frame: Baseline, 18 months up to 24 months
Population: All enrolled participants.
Measure: Number; unit: participants
Arm/Group | Ruboxistaurin
Number analyzed (Participants) | 203
participants | 10 [2 to 9]

2. Secondary Outcome: Vision Loss
Description: The number of participants whose best-corrected Early Treatment Diabetic Retinopathy Study (ETDRS) visual acuity (VA) in at least 1 diabetic retinopathy (DR) study eye decreased by 15-letters or less from the conclusion of Study MBCM to the start of Study MBDV, 6 to 18 months later. Best-corrected ETDRS VA was measured at 4 meters (m) using an eye chart with 5 letters per row of decreasing letter size in each successive row. Participants read the chart from the top down until reaching a row where ≥3 letters in the row could not be read correctly. If <20 letters were read correctly at 4 m, the chart was re-read at 1 m. The best-corrected ETDRS VA score was the total number of letters read correctly per eye at 4 m, plus a correction factor of 30 if ≥20 letters were read correctly at 4 m, plus the total number of letters read correctly at 1 m, if assessed. Best-corrected ETDRS VA scores ranged from 0 (no letters read correctly) to 100 (all letters read correctly).
Time Frame: End of Study MBCM to the beginning of Study MBDV, approximately 6 to 18 months
Population: All enrolled participants.
Measure: Number; unit: participants
Arm/Group | Ruboxistaurin
Number analyzed (Participants) | 203
participants | 22 [7 to 16]

3. Secondary Outcome: Sustained Moderate Vision Loss (SMVL), Long Term
Description: The number of participants who experienced SMVL, long term, in at least 1 diabetic retinopathy (DR) study eye. Long term SMVL was a ≥15-letter decrease from Study MBCM baseline in best-corrected Early Treatment Diabetic Retinopathy Study (ETDRS) visual acuity (VA) that was sustained for the last 6 months of Study MBDV. VA was measured at 4 meters (m) using an eye chart with 5 letters per row of decreasing letter size in each successive row. Participants read the chart from the top down until reaching a row where ≥3 letters in the row could not be read correctly. If <20 letters were read correctly at 4 m, the chart was re-read at 1 m. The best-corrected ETDRS VA score was the total number of letters read correctly per eye at 4 m, plus a correction factor of 30 if ≥20 letters were read correctly at 4 m, plus the total number of letters read correctly at 1 m, if assessed. Best-corrected ETDRS VA scores ranged from 0 (no letters read correctly) to 100 (all letters read correctly).
Time Frame: Baseline in Study MBCM, 18 months up to 24 months in Study MBDV (for a total of 75 up to 87 months of SMVL, long term)
Population: Participants who were treated with 32 milligram (mg) ruboxistaurin once daily in Study MBCM and had at least 1 DR study eye, who were also enrolled in Study MBDV.
Measure: Number; unit: participants
Arm/Group | Ruboxistaurin
Number analyzed (Participants) | 103
participants | 8 [3 to 15]

4. Secondary Outcome: Number of Participants With a Modified Sustained Moderate Vision Loss (mSMVL) Event by Time Interval
Description: An mSMVL event was defined as a ≥15-letter decrease from Study MBDV baseline in best-corrected Early Treatment Diabetic Retinopathy Study (ETDRS) visual acuity (VA) during any 6-month period, not just the last 6 months of the study. An mSMVL event was the first occurrence of an mSMVL in a participant, and the time at which the mSMVL began was used as the time of the event for the analysis. VA was measured at 4 meters (m) using an eye chart with 5 letters per row. Participants read the chart from the top down until reaching a row where ≥3 letters in the row could not be read correctly. If <20 letters were read correctly at 4 m, the chart was re-read at 1 m. The best-corrected ETDRS VA score was the total number of letters read correctly per eye at 4 m, plus a correction factor of 30 if ≥20 letters were read correctly at 4 m, plus the total number of letters read correctly at 1 m, if assessed.
Time Frame: Baseline up to 6 months, 6 months up to 12 months, 12 months up to 18 months, 18 months up to 24 months, and 24 months up to 30 months
Population: All enrolled participants (pts) at risk during the specified intervals. Pts who did not experience an event during the interval were censored to the last time point in the interval. Number of pts censored: 0 to 6 months = 2 pts, 6 to 12 months = 4 pts, 12 to 18 months = 9 pts, 18 to 24 months = 82 pts, and 24 to 30 months = 90 pts.
Measure: Number; unit: participants
Arm/Group | Ruboxistaurin
Number analyzed (Participants) | 198
participants
  0 up to 6 months, n=198 | 0
  6 up to 12 months, n=196 | 4
  12 up to 18 months, n=188 | 5
  18 up to 24 months, n=174 | 2
  24 up to 30 months, n=90 | 0

5. Secondary Outcome: Visual Acuity
Description: Best-corrected Early Treatment Diabetic Retinopathy Study (ETDRS) visual acuity (VA) was measured at 4 meters (m) using an eye chart with 5 letters per row of decreasing letter size in each successive row. Participants read the chart from the top down until reaching a row where ≥3 letters in the row could not be read correctly. If <20 letters were read correctly at 4 m, the chart was re-read at 1 m. The best-corrected ETDRS VA score was the total number of letters read correctly per eye at 4 m, plus a correction factor of 30 if ≥20 letters were read correctly at 4 m, plus the total number of letters read correctly at 1 m, if assessed. Best-corrected ETDRS VA scores ranged from 0 (no letters read correctly) to 100 (all letters read correctly). A higher score represented better VA.
Time Frame: Month 24
Population: All enrolled participants. Last observation carried forward (LOCF).
Measure: Mean (Standard Deviation); unit: letters read correctly
Arm/Group | Ruboxistaurin
Number analyzed (Participants) | 203
letters read correctly | 75.14 (14.92)

6. Secondary Outcome: Number of Participants Receiving Treatment With Focal/Grid Photocoagulation
Time Frame: Baseline up to Month 24
Population: All enrolled participants.
Measure: Number; unit: participants
Arm/Group | Ruboxistaurin
Number analyzed (Participants) | 203
participants | 19 [6 to 14]

7. Secondary Outcome: Number of Participants Receiving Treatment With Panretinal Photocoagulation
Time Frame: Baseline up to Month 24
Population: All enrolled participants.
Measure: Number; unit: participants
Arm/Group | Ruboxistaurin
Number analyzed (Participants) | 203
participants | 53 [20 to 33]

ADVERSE EVENTS:
Arm/Group | Ruboxistaurin
Serious Adverse Events (participants affected / at risk) | 57/203
Other Adverse Events (participants affected / at risk) | 166/203
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ruboxistaurin (N=203)
Anaemia (Blood and lymphatic system disorders) | 1 (1)
Acute myocardial infarction (Cardiac disorders) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (1)
Bradycardia (Cardiac disorders) | 1 (1)
Cardiac arrest (Cardiac disorders) | 1 (2) — Event resulted in 1 death
Cardiac failure congestive (Cardiac disorders) | 8 (15) — Event resulted in 1 death
Cardio-respiratory arrest (Cardiac disorders) | 1 (1) — Event resulted in 1 death
Cardiopulmonary failure (Cardiac disorders) | 1 (1) — Event resulted in 1 death
Coronary artery disease (Cardiac disorders) | 6 (6)
Hypertensive heart disease (Cardiac disorders) | 1 (1)
Ischaemic cardiomyopathy (Cardiac disorders) | 1 (1)
Myocardial infarction (Cardiac disorders) | 2 (2)
Sick sinus syndrome (Cardiac disorders) | 1 (1)
Ventricular dysfunction (Cardiac disorders) | 1 (1)
Ventricular tachycardia (Cardiac disorders) | 1 (1)
Acute abdomen (Gastrointestinal disorders) | 1 (1)
Erosive oesophagitis (Gastrointestinal disorders) | 1 (1)
Gastric ulcer (Gastrointestinal disorders) | 1 (1)
Gastritis (Gastrointestinal disorders) | 1 (1)
Gastritis erosive (Gastrointestinal disorders) | 1 (1)
Impaired gastric emptying (Gastrointestinal disorders) | 1 (1)
Intestinal obstruction (Gastrointestinal disorders) | 2 (2)
Nausea (Gastrointestinal disorders) | 1 (1)
Oesophagitis (Gastrointestinal disorders) | 1 (1)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
Chest pain (General disorders) | 4 (4)
Death (General disorders) | 1 (1)
Generalised oedema (General disorders) | 1 (1)
Oedema peripheral (General disorders) | 1 (1)
Appendicitis (Infections and infestations) | 1 (1)
Arthritis infective (Infections and infestations) | 1 (1)
Bronchitis (Infections and infestations) | 1 (1)
Cellulitis (Infections and infestations) | 7 (8)
Endocarditis (Infections and infestations) | 1 (1)
Gangrene (Infections and infestations) | 1 (1)
Gastroenteritis (Infections and infestations) | 1 (1)
Gastroenteritis viral (Infections and infestations) | 1 (1)
Infection (Infections and infestations) | 1 (1)
Kidney infection (Infections and infestations) | 1 (1)
Localised infection (Infections and infestations) | 1 (1)
Osteomyelitis (Infections and infestations) | 4 (4)
Pneumonia (Infections and infestations) | 4 (4)
Pyelonephritis acute (Infections and infestations) | 1 (1)
Septic shock (Infections and infestations) | 1 (1) — Event resulted in 1 death
Sinusitis (Infections and infestations) | 1 (1)
Staphylococcal abscess (Infections and infestations) | 1 (1)
Staphylococcal bacteraemia (Infections and infestations) | 1 (1)
Urinary tract infection (Infections and infestations) | 3 (3)
Urosepsis (Infections and infestations) | 1 (1)
Viral infection (Infections and infestations) | 1 (1)
Wound infection staphylococcal (Infections and infestations) | 1 (1)
Acetabulum fracture (Injury, poisoning and procedural complications) | 1 (1)
Foot fracture (Injury, poisoning and procedural complications) | 1 (1)
Hip fracture (Injury, poisoning and procedural complications) | 1 (1)
Lower limb fracture (Injury, poisoning and procedural complications) | 1 (1)
Pocket erosion (Injury, poisoning and procedural complications) | 1 (1)
Rib fracture (Injury, poisoning and procedural complications) | 1 (1)
Subdural haematoma (Injury, poisoning and procedural complications) | 1 (1)
Heart rate irregular (Investigations) | 2 (2)
Dehydration (Metabolism and nutrition disorders) | 3 (3)
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) — Event resulted in 1 death
Fistula (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1)
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Brain stem infarction (Nervous system disorders) | 1 (1)
Carotid artery occlusion (Nervous system disorders) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 1 (1)
Cervicobrachial syndrome (Nervous system disorders) | 1 (1)
Coma (Nervous system disorders) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1)
Syncope (Nervous system disorders) | 3 (3)
Transient ischaemic attack (Nervous system disorders) | 2 (2)
Diabetic nephropathy (Renal and urinary disorders) | 1 (1)
Renal failure acute (Renal and urinary disorders) | 6 (6) — Event resulted in 1 death
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Event resulted in 1 death
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 3 (4)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1)
Toe amputation (Surgical and medical procedures) | 1 (1)
Arteriosclerosis (Vascular disorders) | 1 (1)
Hypertensive emergency (Vascular disorders) | 1 (1)
Hypotension (Vascular disorders) | 2 (2)
Malignant hypertension (Vascular disorders) | 1 (1)
Orthostatic hypotension (Vascular disorders) | 1 (1)
Peripheral vascular disorder (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ruboxistaurin (N=203)
Vitreous haemorrhage (Eye disorders) | 20 (25)
Diarrhoea (Gastrointestinal disorders) | 16 (19)
Bronchitis (Infections and infestations) | 12 (14)
Nasopharyngitis (Infections and infestations) | 22 (32)
Upper respiratory tract infection (Infections and infestations) | 11 (11)
Urinary tract infection (Infections and infestations) | 13 (21)
Back pain (Musculoskeletal and connective tissue disorders) | 18 (20)
Cough (Respiratory, thoracic and mediastinal disorders) | 15 (19)
Cataract operation (Surgical and medical procedures) | 15 (20)
Retinal laser coagulation (Surgical and medical procedures) | 49 (111)
Vitrectomy (Surgical and medical procedures) | 12 (16)

LIMITATIONS AND CAVEATS:
A participant could have one or both eyes meet the criteria for a diabetic retinopathy (DR) study eye as defined in study B7A-MC-MBCM.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days